CLINICAL TRIAL: NCT06960967
Title: Postprandial Effects of Chestnuts on Glycaemic Response: a Cross-over Trial in Healthy Adults
Brief Title: Effects of Chestnuts on Postprandial Glycaemic Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbara R. Cardoso, PhD, Monash University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ChestnutsProject
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Postprandial Glycemia; Insulin Resistance
Keywords: chestnuts; postprandial glycemia; postprandial insulinemia; glucose tolerance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The participants will be requested to attend 2 morning visits to the research centre to receive one of the test meals. These meals will be isocaloric with or without the addition of chestnut flour. The order in which they undertake the two test visits will be randomised.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control meal (Placebo Comparator): Participants will receive an isocaloric baked meal without chestnut flour.
  Interventions: Other: Control meal
- Chestnut meal (Experimental): Participants will receive an isocaloric baked meal with chestnut flour.
  Interventions: Other: Chestnut meal

INTERVENTIONS:
Other: Chestnut meal — Participants will receive an isocaloric baked meal with chestnut flour.
  Arms: Chestnut meal
Other: Control meal — Participants will receive an isocaloric baked meal without chestnut flour.
  Arms: Control meal

SUMMARY:
Nut consumption is known to improve health outcomes, such as reducing the risk of chronic diseases like diabetes, cognitive impairment, and cardiovascular diseases. While most research has focused on walnuts and almonds, there is limited information on the health benefits of chestnuts. Chestnuts are unique among tree nuts due to their high starch and fibre content, along with vitamins E and C, minerals (potassium, phosphorus, magnesium), and polyphenols.

Evidence from in vitro and animal studies suggests that chestnuts may positively affect health by regulating the gut microbiome, lowering the glycaemic index, and providing antioxidant benefits. The food industry is also exploring new uses for chestnuts, particularly in gluten-free products, due to their nutritional benefits and good taste. Nonetheless, no research has investigated the health effects of chestnuts in humans. By addressing this gap in the literature, the study may lead to the development of new dietary strategies for improved health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years old
* Available to attend two testing sessions at the research facility

Exclusion Criteria:

* Allergy to nuts and/or gluten,
* BMI<18.5 or ≥30 kg/m2,
* Fasting glucose >5.6 mmol/L, presence of diabetes and/or taking anti-diabetic medication
* Serious health conditions that may affect participation e.g. liver or thyroid dysfunction, recent major surgery,
* Smoker,
* Cardiovascular disease
* Pregnant or breastfeeding women
* Presence of implanted cardiac defibrillator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Postprandial blood glucose incremental area under the curve (iAUC) | Three hour blood glucose iAUC will be calculated from nine time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial blood glucose iAUC
Postprandial plasma insulin incremental area under the curve (iAUC) | Three hour insulin iAUC will be calculated from seven time points (0, 30, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial plasma insulin iAUC.

SECONDARY OUTCOMES:
Postprandial glucose concentration | Glucose concentration will be measured at nine time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial glucose concentration
Postprandial insulin concentration | Insulin concentration will be measured in finger prick blood samples at seven time points (0, 30, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial insulin concentration
Time to peak glucose | Three hours
  Difference in time to peak glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No